CLINICAL TRIAL: NCT00964145
Title: Effects of Age on the Levator Ani Muscle of Nulliparous Women
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Lieschen H. Quiroz, M.D., University of Oklahoma Health Sciences Center
Other Study IDs: 14723 Nulliparous Women
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Nulliparous Women
Keywords: Nulliparous women; ultrasound

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nulliparous female patients: Nulliparous female patients ages 21-70 years old.

SUMMARY:
The purpose of the study is to characterize the levator ani structures (pubovaginalis, puboperinealis, puboanalis, puborectalis, and the iliococcygeous) using 3-D ultrasonography in nulliparous women 21-70 years old.

Hypothesis 1: Prevalence of abnormalities in levator ani muscle structure will be associated with increasing age independent of vaginal parity. To investigate the age-related symptoms of pelvic floor dysfunction in nulliparous, women 21-70 years old.

Hypothesis 2: Anatomical abnormalities of the levator ani muscles will be associated with symptomatic pelvic floor dysfunction. To investigate the age-related pelvic floor function in nulliparous, women 21-70 years old.

Hypothesis 3: Age-related anatomical abnormalities of the levator ani muscles will be associated with levator ani muscle weakness.

DETAILED DESCRIPTION:
This is a a cross-sectional study of age-related changes in the levator ani muscles. We will explore the 3-D anatomical architecture of these muscles in asymptomatic females ages 21-70 years old. Subjects who meet eligibility criteria will be scheduled to have a clinic study visit during which informed consent will be obtained. At this visit, subjects will be asked to complete self administered pelvic floor symptom and impact measures questionnaire (PFDI, PFIQ and PISQ-12), as well as the quality of life measure (SF-12). At the clinic study visit, a complete history will be obtained including the subject's gynecologic history including age, menopausal status, medical and surgical history by interview. A standardized examination will performed, including height, weight, and pelvic floor support assessment by using the pelvic organ prolapse quantification system (POP-Q). Body mass index will be calculated. Levator function will be assessed using the instrumented vaginal speculum. Vaginal closure force will be measured at both rest and during maximal voluntary contraction. At the completion of the exam and speculum examinations, all participants will then undergo an endovaginal 3-D ultrasound (BK medical, Wilmington, MA), at the study visit. The endovaginal ultrasound technique has been described previously. The technique is summarized as follows: A length of six cm will be scanned in 60 seconds at scans every 0.25 mm with a cumulative 240 scans from which a 3-D rendered cube will be calculated. Each 3-D cube will be digitally catalogued for future analysis. The ultrasound cubes will then be reviewed by two reviewers (LHQ and SAS), blinded to the identity of volunteers or the scores of the other reviewer. Reviewers will score muscles based on the individual muscle visualization by the origin - insertion points. The levator ani muscles in these scans will be examined for the visibility of the puboperinealis, puboanalis and pubovaginalis divisions of the levator ani muscle. Other structures, such as the superficial transverse perinei, puborectalis and iliococcygeous muscle will also be identified. A scoring system was previously developed according to the morphology and clarity of the each subdivision's origin-insertion points. The characteristic features of each levator subdivision will determined by the following two criteria: A clear and visible separation between each adjacent structure, or, Differing origin-insertion points of the muscle. An exemplary scan of a 25 year-old nulliparous women has been selected for image clarity based on the described classification method. According to the scoring system, a score of 0 given to each muscle pair corresponds to "no muscle damage" and a score of 18 corresponds to "complete muscle loss" of all subdivisions. Next, a 3-D PowerPoint library will be created describing the structures that need to be identified. The blinded reviewer may confirm the identity of the structure by manipulating the planes on the 3-D cube to trace the entire muscle subdivision to look for origin-insertion points.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous female patients ages 21-70 years old

Exclusion Criteria:

* History of prior incontinence, or prolapse surgery
* Diagnosis of reproductive tract anomalies
* Prior pelvic radiation therapy
* Hysterectomy
* Unable to complete written questionnaires

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling nulliparous females, ages 21-70 years. Women are eligible for participation if they are willing to undergo a physical examination regardless of race, continence or prolapse status.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To characterize the levator ani structures (pubovaginalis, puboperinealis, puboanalis, puborectalis, and the iliococcygeous) using 3-D ultrasonography in nulliparous women 21-70 years old. | August 2011
To investigate the age-related pelvic floor dysfunction in nulliparous women 21-70 years old. | August 2011
To investigate the age-related pelvic floor function in nulliparous, women 21-70 years old. | August 2011

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen H. Quiroz, M.D., Principal Investigator — University of Oklahoma Health Sciences Center/Medicine/OB/GYN
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States